CLINICAL TRIAL: NCT05149950
Title: Internet Treatment for Patients With Obesity - a Randomized Study
Brief Title: Internet Treatment for Patients With Obesity
Acronym: ROLobes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Örebro County (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 276484
Record Dates: First submitted 2021-11-03; First posted 2021-12-08 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Increased therapist contact. (Experimental): The patient gets access to the internet treatment via a secure login to 1177 The care guide-services on 1177.se. The treatment lasts for six months and includes 12 treatment modules. The patient works with each module for two weeks. The modules have different numbers of sections, but most have 4-5 sections. The modules consist mainly of text but also films and pictures are included. It is also possible to listen to the text. The modules end with one or more exercises to be performed before the next module is activated for the patient. Participants receive feedback on the information from therapists via the email function in the treatment program. The therapist provides individual feedback on completed exercises and answers questions that the patient has.
  Interventions: Behavioral: Active internet treatment
- Less therapist contact. (Other): The feedback from the therapist will largely be general and not individually tailored. The general feedback is based on responses to the participants in the previous pilot study. No physical or digital meetings between patient and therapist take place during treatment.
  Interventions: Behavioral: Active internet treatment

INTERVENTIONS:
Behavioral: Active internet treatment — The patient gets access to the internet treatment via a secure login to 1177 The care guide e-services on 1177.se. The treatment lasts for six months and includes 12 treatment modules. The patient works with each module for two weeks. The modules have different numbers of sections, but most have 4-5 sections. The modules consist mainly of text but also films and pictures are included. It is also possible to listen to the text. The modules end with one or more exercises to be performed before the next module is activated for the patient. Participants receive feedback on the information from therapists via the email function in the treatment program. The therapist provides individual feedback on completed exercises and answers questions that the patient has.

SUMMARY:
There is a strong link between obesity and reduced quality of life as well as serious sequelae of diseases. Step by step is a treatment model that has been developed at the Obesity Unit, Orebro County Region and includes six group meetings over 6-8 months. The aim is to increase patients' knowledge about the disease obesity, to provide support for lifestyle changes and weight control, and to reduce stigma-related psychosocial disorders. A 1-year pilot study aimed at evaluating the Internet-based Step by Step treatment has recently been completed. Results after 6 months of treatment show that the participants who completed the treatment were mainly satisfied with the program and the content. However, the dropouts from the treatment were more than expected.

DETAILED DESCRIPTION:
Based on the experience from the pilot study, a new randomized study is planned with the aim of evaluating a revised treatment program. People 25-69 years with a BMI 30-44.9 kg / m2, or with a BMI 28-29.9 kg / m2 and co-occurrence of hypertension, prediabetes, type 2 diabetes, coronary heart disease, hyperlipidemia, hepatic steatosis, sleep apnea or polycystic ovary syndrome can be included. The intervention group receives increased therapist support with physical or digital meetings before and during the treatment as well as individualized feedback from the therapist. Feedback takes place after 6, 12 and 18 weeks. The other group, the control group, implements the program without meetings with the therapist and receives general feedback during the treatment. The purpose is to evaluate whether increased therapist contact compared to less therapist contact leads to improved weight reduction, quality of life, eating habits and increases physical activity at follow-up after 12 months

ELIGIBILITY:
Inclusion Criteria:

* BMI 30-44.9 kg / m2
* BMI 28-29.9 kg / m2 and hypertension
* BMI 28-29.9 kg / m2 and prediabetes
* BMI 28-29.9 kg / m2 and type 2 diabetes
* BMI 28-29.9 kg / m2 and coronary heart disease
* BMI 28-29.9 kg / m2 and hyperlipidemia
* BMI 28-29.9 kg / m2 and hepatic steatosis
* BMI 28-29.9 kg / m2 and sleep apnea
* BMI 28-29.9 kg / m2 and polycystic ovary syndrome

Exclusion Criteria:

* Severe mental illness
* Ongoing or suspected eating disorder
* Pregnancy
* Breastfeeding
* Cancer in active treatment
* Use of drugs for weight loss
* Weight loss treatment during the past 6 months
* Active abuse of alcohol or drugs
* Not being able to express themselves in Swedish in speech and writing
* If the study supervisor deems that participation in the study is inappropriate for another reason.

Ages: 25 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-01-03 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Obesity-specific quality of life | 12 months
  Avoidant social behavior due to obesity-related psychosocial disorders which is measured with the Obesity-related Problems scale "(OP)". The OP scale is validated to measure obesity-specific quality of life. OP measures the negative effects of obesity on psychosocial functioning and is useful for evaluating the effects of obesity interventions on quality of life. Scores range from 0 to 100, and higher scores indicate dysfunction.

SECONDARY OUTCOMES:
Weight reduction as a percentage of body weight before treatment | 6 and 12 months
  Each participant's weight reduction in kilograms reported as a percentage of body weight before starting treatment
Proportion of participants with ≥ 5% weight reduction | 6 and 12 months
  Proportion of participants with ≥ 5% weight reduction in kilograms
General health-related quality of life | 6 and 12 months
  General quality of life is measured with RAND-36 which consists of 36 questions and measures 8 health domains: physical function, role function-physical, pain, general health, energy / fatigue, social function, role function-emotional and emotional well-being. Using the standard scoring algorithm from RAND Corporation, eight conceptual attributes (subscales) are calculated by averaging values of 35 of the 36 ordinal scale items. The remaining item (general health change), assesses change in perceived health during the last year. Subscale scores range from 0 to 100, where higher scores represent better health status.The Swedish version is validated
Obesity-specific quality of life: psychosocial distress | 6 and 12 months
  Psychosocial distress due to obesity-related problems is measured with the Obesity-related Problems scale "(OP)". The OP scale is validated to measure obesity-specific quality of life. OP measures the negative effects of obesity on psychosocial functioning and is useful for evaluating the effects of obesity interventions on quality of life. Scores range from 0 to 100, and higher scores indicate dysfunction.
Dietary habits | 6 and 12 months
  Dietary habits are measured by the National Board of Health and Welfare's five dietary index questions. The questions measure how often the person eats 1) vegetables, 2) fruit, 3) fish, 4) coffee bread / chocolate / sweets / soft drinks, and 5) how often the person eats breakfast.
Physical activity | 6 and 12 months
  Measured with the National Board of Health and Welfare three indicator questions about exercise, exercise and sitting still. The questions measure how much time per week the person performs 1) strenuous activities, e.g. running, playing ball, and 2) moderately strenuous activities, e.g. walking, cycling and 3) how many hours during the day the person is sedentary.
Physical activity measured with an accelerometer | During 7 days before treatment and at 6 and 12 months
  Measured with an accelerometer for 7 days before treatment and at follow-up at 6 and 12 months after the start of treatment. The measurement is made with the Actigraph GTX3 + monitor which is distributed or sent home to participants at the above times. Data on physical activity are combined with body weight to calculate energy consumption. During the 7 days that the survey takes place, the participants document various activities in a diary.
Eating behavior | 6 and 12 months
  Eating behavior is measured with the Three-Factor Eating Questionnaire-Revised 18 items (TFEQ-R18v2) which is a validated questionnaire consisting of 18 questions that measure three aspects of eating behavior: uncontrolled eating (tendency to lose control over intake when you feel hungry or when you exposed to external stimuli), cognitive restraint (conscious restriction of food intake to control body weight or body shape) and emotional eating (overeating in connection with negative emotional states).Responses are scored on a 4-point scale, and anchors can vary across items (e.g., definitely true to definitely false, or never to at least once a week). Means are computed for each subscale (as long as at least half of the items have been answered) and are transformed to correspond to a 0-100 scale score. A higher score indicates more restraint, uncontrolled, and emotional eating.
Sleep quality | 6 and 12 months
  Measured with the Insomnia Severity Index (ISI) which consists of 7 questions that evaluate sleep, sleep during the night, waking up early, the feeling of being rested, how the sleep problems affect daily life, and whether the sleep pattern worries the individual. The scale score ranges between 0-28 and a higher score indicates more sleep problems.
Completion of the treatment program | 6 and 12 months
  Percentage who complete the treatment program
The participants' experiences and experiences of the treatment | Every three weeks up to 24 weeks
  The patient's experience of the treatment program is measured with questions after each treatment module and at the end of treatment after 6 months. The questionnaire questions are answered in the treatment platform and contain questions about:
  * how easy or difficult it is to follow the treatment program
    * to understand the language
    * to absorb the content
    * to access and use the program
    * to understand the homework and whether these were relevant / helpful
    * how helpful the feedback from the therapist is
    * what can be improved

CONTACTS AND LOCATIONS:
Overall Officials: Mats G Karlsson, Prof, Study Chair — Region Orebro County
Locations (1):
- Stefan Jansson, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No